CLINICAL TRIAL: NCT05980975
Title: The Effect of Coffee and Hot Water Consumptıon on Gastroıntestınal System Functıons After Cesarrean Sectıon
Brief Title: The Effect of Coffee and Hot Water on Gastroıntestınal Functıons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Seher Gürdil Yılmaz, Lecturer doctor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinUniversityy
Record Dates: First submitted 2023-07-14; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: COFFEE; Gastrointestinal Motility and Defecation Conditions
Keywords: cesarean section; coffee; bowel sound; flatulence
MeSH Terms: conditions — Flatulence | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coffee group (Group 1) (Experimental): Then, at the 4th hour, 8th hour and 12th hour of the surgery, the patients in the coffee group received 10 gr. granulated coffee.
  Interventions: Other: Coffee
- Hot water group (Group 2) (Experimental): The patients in the hot water group were given 200 ml of 50-60 C0 sugar-free hot water at the 4th hour, 8th hour and 12th hour of the operation.
  Interventions: Other: Hot water
- Control group (Group 3) (No Intervention): No application was made to the control group.

INTERVENTIONS:
Other: Coffee — 4th hour, 8th hour and 12th hour of after the surgery, the patients in the coffee group received 10 gr. granulated coffee.
  Arms: Coffee group (Group 1)
Other: Hot water — hot water group were given 200 ml of 50-60 C0 sugar-free hot water at the 4th hour, 8th hour and 12th hour of after the operation
  Arms: Hot water group (Group 2)

SUMMARY:
The aim of this study is to examine the effects of coffee and hot water consumption on gastrointestinal system functions after cesarean section performed under general anesthesia. The study is in a randomized controlled experimental design.

The sample of the study consisted of 25 participants in the coffee group (Group 1), 26 participants in the hot water group (Group 2) and 27 participants in the control group (Group 3). After cesarean section, at the 4th, 8th and 12th hours of the operation, the first intervention group (coffee group) received 2 gr. granulated coffee, the second intervention group (hot water group) was given 100 ml of 50-60 C0 sugar-free hot water, the third group (control group) was given no intervention other than routine applications.

DETAILED DESCRIPTION:
Objective: The aim of this study is to examine the effects of coffee and hot water consumption on gastrointestinal system functions after cesarean section performed under general anesthesia.

Materials and Methods: The study is in a randomized controlled experimental design. Patients who had an uncomplicated cesarean section under general anesthesia, were older than 18 years of age, completed the 37th week of pregnancy, did not have any gastrointestinal system disease that could affect the results of the study, and did not use drugs, and who could understand and speak Turkish were included in the study. The sample of the study consisted of 25 participants in the coffee group (Group 1), 26 participants in the hot water group (Group 2) and 27 participants in the control group (Group 3). After cesarean section, at the 4th, 8th and 12th hours of the operation, the first intervention group (coffee group) received 2 gr. granulated coffee, the second intervention group (hot water group) was given 100 ml of 50-60 C0 sugar-free hot water, the third group (control group) was given no intervention other than routine applications.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section performed by the physician determined in the research
* Over 18 years old,
* Completing the 37. gestational week,
* Do not have any gastrointestinal system disease that may affect the results of the research and do not use drugs,
* Able to understand and speak Turkish,
* Women who voluntarily participated in the study

Exclusion Criteria:

* Cesarean section performed by a different physician than the physician determined in the study.
* Younger than 18,
* Not completing the 37.gestational week
* Having any gastrointestinal system disease that may affect the research results and using medication
* Can't understand or speak Turkish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cesarean section is performed only on women.
Enrollment: 77 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
First bowel sound time listened with stethoscope | 24 hours
  After cesarean section, the four quadrants of the abdomen were listened to every hour for the first 12 hours and every 4 hours for the next 12 hours by the investigator, and the first bowel sound time was determined by the investigator.
First gas output, first defecation output, nausea and vomiting by the patient's statement checklist | 24 hours
  Nausea, vomiting, first gas and first defecation times were determined by the patient's statement.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)